CLINICAL TRIAL: NCT00049244
Title: A Phase I Study of BMS-247550 in Combination With Capecitabine in Patients With Metastatic Breast Cancer Previously Treated With a Taxane and an Anthracycline
Brief Title: BMS-247550 Plus Capecitabine in Treating Patients With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: R-Pharm (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: BMS-CA163-031; UCLA-0206011; CDR0000258052 (Registry Identifier: PDQ (Physician Data Query)); NCI-G02-2120
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; ixabepilone

INTERVENTIONS:
Drug: capecitabine
Drug: ixabepilone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining BMS-247550 with capecitabine in treating patients who have metastatic breast cancer that has not responded to previous chemotherapy with a taxane and an anthracycline.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of BMS-247550 and capecitabine, on 2 different schedules, in patients with metastatic breast cancer previously treated with a taxane and an anthracycline.
* Determine the safety profile of this regimen in these patients.
* Determine, preliminarily, any antitumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 2 groups.

* Group I: Patients receive BMS-247550 IV over 3 hours on day 1 and oral capecitabine twice daily on days 1-14.
* Group II: Patients receive BMS-247550 IV over 1 hour on days 1-3 and capecitabine as in group I.

Treatment in both groups repeats every 3 weeks for 2-18 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of BMS-247550 and capecitabine until the maximum tolerated dose (MTD) is determined for each group. The MTD is defined as the dose at which no more than 1 of 6 patients experiences dose-limiting toxicity. Additional patients are treated at the MTD.

Patients are followed for at least 30 days and then every 3 months thereafter.

PROJECTED ACCRUAL: Approximately 34-60 patients will be accrued for this study within 8-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Metastatic disease by radiography or histology
* Must have received prior chemotherapy with a taxane and an anthracycline in the adjuvant or metastatic setting

  * No more than 2 prior chemotherapy regimens in the metastatic setting
* Measurable or evaluable disease

  * Bone lesions not measurable
  * Primary breast lesions not measurable if assessed only by physical exam
* No active brain metastasis

  * No cerebral edema by CT scan or MRI
  * No progression since prior imaging studies
  * No requirement for steroids
  * No clinical symptoms of brain metastasis
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Not specified

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT no greater than 2.5 times ULN

Renal

* Creatinine less than 1.5 times ULN

Cardiovascular

* No uncontrolled or significant cardiovascular disease
* No myocardial infarction within the past year
* No uncontrolled angina within the past year
* No history of congestive heart failure
* No history of atrial or ventricular arrhythmias
* No history of second- or third-degree heart block
* No uncontrolled hypertension

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No hypersensitivity to Cremophor EL or fluorouracil
* No prior intolerance to fluoropyrimidines
* No other serious uncontrolled medical disorder or active infection that would preclude study
* No dementia or altered mental status that would preclude study
* No grade 2 or greater neuropathy (neuromotor or neurosensory)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Chemotherapy
* Prior immunotherapy allowed
* No concurrent trastuzumab (Herceptin)
* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas, mitomycin, or doxorubicin HCl liposome)
* At least 2 years since prior high-dose chemotherapy with bone marrow transplantation or peripheral blood stem cell support
* No prior epothilone, capecitabine, or continuous-infusion fluorouracil
* No other concurrent chemotherapy

Endocrine therapy

* Prior hormonal therapy allowed
* No concurrent hormonal therapy
* Concurrent hormone replacement therapy allowed

Radiotherapy

* At least 3 weeks since prior radiotherapy
* No prior radiotherapy to more than 25% of the bone marrow
* No concurrent therapeutic radiotherapy

Surgery

* Not specified

Other

* At least 3 weeks since prior investigational cytotoxic agents
* No concurrent warfarin for therapeutic anticoagulation

  * Low-dose warfarin allowed for implanted ports or indwelling catheters
* No other concurrent experimental anticancer medications
* No other concurrent antitumor therapy
* Concurrent bisphosphonates for palliation of bone metastases allowed if initiated before study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Linnea Chap, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States